CLINICAL TRIAL: NCT01325623
Title: Seizure Detection and Automatic Magnet Mode Performance Study
Acronym: E-36
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cyberonics, Inc. (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Epilepsy (E)-36
Record Dates: First submitted 2011-03-23; First posted 2011-03-30 (Estimated); Results first posted 2016-01-22 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2015-12

CONDITIONS: Epilepsy
Keywords: Automatic Magnet Mode (AMM); Vagal Nerve Stimulation
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Model 106 VNS Therapy System (Other): Model 106 VNS Therapy System includes a new Seizure Detection Algorithm (SDA) and corresponding Automatic Magnet Mode (AMM) feature.
  Interventions: Device: Model 106 VNS Therapy System

INTERVENTIONS:
Device: Model 106 VNS Therapy System — The VNS Therapy System is an adjunctive therapy for the treatment of epilepsy. VNS Therapy is available as a scheduled stimulation, this is cyclic stimulation between programmable On- and Off- times (e.g., a 30-second burst every 5 minutes). VNS Therapy is also available as on-demand stimulation, that is, when a magnet is introduced briefly over the implanted device (Magnet Mode). The AspireSR VNS Therapy System includes a new feature, Automatic Magnet Mode or AutoStim. In addition to Normal Mode and Magnet Mode, AspireSR uses a Seizure Detection Algorithm to identify a potential seizure onset based on associated heart rate increases known as ictal tachycardia. The purpose is to deliver stimulation at or near the onset of a seizure.
  Other Names: AspireSR VNS Therapy System

SUMMARY:
The purpose of this study is to confirm cardiac-based seizure detection in Cyberonics Model 106 VNS Therapy System.

DETAILED DESCRIPTION:
Prospective, observational, unblinded, multi-site study designed to collect data on patients implanted with a Model 106 VNS Therapy System from baseline through an EMU stay of up to 5 days. After the EMU stay, patients will continue follow-up for safety for approximately two years or until final regulatory approval of the product.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of medically refractory epilepsy dominated by partial seizures suitable for implantation with the Model 106 VNS Therapy System.
* Patients with a history of increased heart rate (tachycardia) associated with seizure onset based on clinical data obtained from medical history, admission/hospital charts, or prior neurophysiologic evaluations.
* Patients willing to undergo an EMU evaluation for a period of at least three days with activation of the AMM feature during that time.
* Patients having an average of ≥ 3 seizures per month based upon diary or patient reporting for the 3 months prior to the screening visit.
* Patients must have peak-peak R-wave amplitude greater than or equal to 0.40 mV on ECG measured from the proposed electrode location in the neck to the proposed generator location in the chest via surface ECG electrodes in 7 different body positions.
* Patients must be at least 18 years old.
* Patients must be in good general health and ambulatory.
* Patient must be willing and able to complete informed consent.

Exclusion Criteria:

* Patients have had a bilateral or left cervical vagotomy.
* Patients currently use, or are expected to use, short-wave diathermy, microwave diathermy, or therapeutic ultrasound diathermy.
* A VNS Therapy System implant would (in the investigator's judgment) pose an unacceptable surgical or medical risk for the patient.
* Patients expected to require full body magnetic resonance imaging.
* Patients have a history of VNS Therapy.
* Patients have a documented history of clinically meaningful bradycardia (heart rate less than 50 bpm) associated with seizures.
* Patients with a significant psychiatric disorder, significant cognitive impairment, history of major depression, or suicidality as defined by DSM IV-TR that in the investigator's judgment would pose an unacceptable risk for the patient or prevent the patient's successful completion of the study.
* Patients with a history of status epilepticus within 3 months of study enrollment.
* Patients prescribed drugs specifically for a cardiac or autonomic disorder that in the investigator's opinion would affect heart rate response unless the patient has ictal tachycardia while taking said drugs. These include, but are not limited to, beta adrenergic antagonists ("beta blockers").
* Patients with known clinically meaningful cardiovascular arrhythmias as well as patients with clinically meaningful cardiovascular arrhythmias determined by a 24-hour Holter recording obtained at the screening visit.
* Patients dependent on alcohol or narcotic drugs as defined by DSM IV-TR within the past 2 years.
* Patients with a history of only psychogenic or pseudo seizures.
* Women who are pregnant. Women of childbearing age must take a pregnancy test.
* Patients currently enrolled in another investigational study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-03; Primary Completion 2013-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Olin, Study Director — Cyberonics, Inc.; Paul Boon, Principal Investigator — University Ghent
Locations (14):
- Belgium (3):
  - Hôpital Erasme, Anderlecht
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
- Germany (6):
  - Epilepsie-Zentrum Bethel, Bielefeld
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Erlangen, Erlangen
  - Albert-Ludwigs-Universität, Freiburg im Breisgau
  - Ludwig-Maximilians-Universität München, Munich
  - Universitätsklinikum Tübingen, Tübingen
- Kempenhaege, Heeze, Netherlands
- Oslo University Hospital, Oslo, Norway
- United Kingdom (3):
  - King's College Hospital, London
  - The National Hospital for Neurology and Neurosurgery, London
  - Royal Hallamshire Hospital, Sheffield

REFERENCES:
- [Result] Boon P, Vonck K, van Rijckevorsel K, El Tahry R, Elger CE, Mullatti N, Schulze-Bonhage A, Wagner L, Diehl B, Hamer H, Reuber M, Kostov H, Legros B, Noachtar S, Weber YG, Coenen VA, Rooijakkers H, Schijns OE, Selway R, Van Roost D, Eggleston KS, Van Grunderbeek W, Jayewardene AK, McGuire RM. A prospective, multicenter study of cardiac-based seizure detection to activate vagus nerve stimulation. Seizure. 2015 Nov;32:52-61. doi: 10.1016/j.seizure.2015.08.011. Epub 2015 Sep 21. PMID 26552564
- [Derived] Verrier RL, Nearing BD, Olin B, Boon P, Schachter SC. Baseline elevation and reduction in cardiac electrical instability assessed by quantitative T-wave alternans in patients with drug-resistant epilepsy treated with vagus nerve stimulation in the AspireSR E-36 trial. Epilepsy Behav. 2016 Sep;62:85-9. doi: 10.1016/j.yebeh.2016.06.016. Epub 2016 Jul 21. PMID 27450311

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible subjects were at least 18 years old, with a clinical diagnosis of medically refractory epilepsy dominated by partial seizures suitable for implantation with the Model 106 VNS Therapy System and a history of ictal tachycardia, defined as heart rate above 100 bpm during a seizure and at least a 55% increase or 35 bpm increase from baseline.
Pre-assignment Details: A total of 35 subjects were screened; (4) did not meet study criteria, (31) were treated/implanted with the AspireSR® VNS Therapy® System, of which (1) was implanted with version 1 of the AspireSR® VNS Therapy® System and (30) were implanted with version 2 (= ITT population).
Groups:
- Enrolled and Treated Population (Safety Population): Consists of all patients who provided consent and were implanted with the AspireSR VNS Therapy System version 1 or version 2. The safety population will be used for all safety analyses. (N=31 subjects).
  In version 2 of the AspireSR VNS Therapy System, the TVS diodes (present in version 1) were removed from the electrical circuit to address the accumulation of electrical charge on the sensing node (e.g. generator-can) following delivery of a stimulation.
Period: Overall Study
Arm/Group | Enrolled and Treated Population (Safety Population)
Started | 31
Completed | 28
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: Subjects who provided consent and were implanted with the AspireSR VNS Therapy System version 1 or version 2.
Groups:
- VNS Therapy (Safety Population): The safety population consists of all patients who provided consent and were implanted with the AspireSR VNS Therapy System version 1 or version 2.
Arm/Group | VNS Therapy (Safety Population)
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (13.4)
Age, Customized [Median (Full Range); unit: years] | 38 [19 to 66]
Age, Customized [Number; unit: participants]
  18-29 years | 10
  30-39 years | 8
  40-49 years | 5
  50-59 years | 5
  60 years or older | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 12
Race/Ethnicity, Customized [Number; unit: participants]
  White | 31
  Other | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 3
  Belgium | 10
  Norway | 1
  United Kingdom | 7
  Germany | 10
Cognitive Status [Number; unit: participants]
  Normal | 20
  Minimal Impairment | 8
  Moderate Impairment | 3
  Severe Impairment | 0
Age at Epilepsy Onset [Median (Full Range); unit: years] | 14 [2 to 43]
Age at Epilepsy Onset [Mean (Standard Deviation); unit: years] | 15.9 (10.9)
Previous Brain or Epilepsy Surgery [Number; unit: participants]
  No | 22
  Yes | 9
Etiology [Number; unit: participants]
  Idiopathic | 3
  Symptomatic | 16
  Cryptogenic | 12
Family History of Seizures [Number; unit: participants]
  No | 24
  Yes | 7
Seizures with Auras in the Past 2 Months [Number; unit: participants]
  No | 15
  Yes | 16

OUTCOME MEASURES:

1. Primary Outcome: Summary of Seizures Reported by Investigators and Triple Review
Description: Subjects were admitted to the EMU and underwent standard continuous data collection of vEEG and ECG for 3 to 5 days. If a seizure occurred during the EMU stay, clinical investigators annotated the start and stop times, the type of seizure, the presumed seizure onset location, and the lobe of origin as applicable.
  Following the EMU data collection phase of the trial, the de-identified, continuous electronic records (per patient) from the EMU period were provided to an independent and blinded triple review panel. This panel evaluated the EEG data and annotated seizure onset, seizure offset, and a description of seizure type. In the absence of video, seizure types could only be specified as: partial (particular type not denoted), generalized (non-absence), absence, or partial with secondary generalization.
Time Frame: Epilepsy Monitoring Unit Stay
Population: ITT Population: consists of all patients implanted with the AspireSR VNS Therapy System version 2 and who have any EMU record.
Measure: Number; unit: Seizures
Groups:
- Reported by Investigators: All seizures that occurred during EMU stay and that were identified by investigators.
- Reported by Triple Review: All seizures that occurred during EMU stay and that were identified by triple review post EMU.
- Total: Seizures from an ITT subject that were either identified by the investigator during EMU evaluation or during the triple review process of EEG data.
Arm/Group | Reported by Investigators | Reported by Triple Review | Total
Number analyzed (Participants) | 30 | 30 | 30
Seizures
  All Seizure Types | 87 | 124 | 211
  Total Partial | 82 | 51 | 133
  Partial | 8 | 51 | 59
  Simple Partial | 26 | 0 | 26
  Complex Partial | 31 | 0 | 31
  Complex Partial with Secondary Generalization | 17 | 0 | 17
  Primary Generalized | 0 | 43 | 43
  Sub-Clinical | 1 | 0 | 1
  Unknown | 3 | 0 | 3
  Other | 1 | 0 | 1
  Unclassified Seizure | 0 | 30 | 30

2. Primary Outcome: Observed Sensitivity Based on Heart Rate Increase Associated With Seizures by Randomized SDA Setting
Description: Sensitivity is the total number of seizures detected divided by the total number of seizures during EMU stay.Data used to support sensitivity analyses included digital ECG/EEG files,corresponding M106 device downloads,and CRF data.Seizure and non-seizure EEG segments were provided to independent reviewers to confirm seizure occurrence and define EEG seizure onset times.Seizure onset times were then compared with observed M106 device detections at the detection threshold setting for AutoStim that the patient was randomized to(SDA 2;60%,SDA 4;40%,SDA 6;20%).Sensitivity is only reported if the heart rate surpassed the programmed detection threshold.Number of participants is total number of subjects who had seizures during the EMU stay.
  An "Ictal tachycardia Seizure" is a seizure with Ictal Heart rate >= 100 bpm & at least 55% increase, or 35 bpm increase from baseline) Bootstrap confidence intervals using 3000 bootstrap samples. n=total number of seizures; N= number of participants
Time Frame: Epilepsy Monitoring Unit (EMU) Stay
Population: Patients from the ITT population who completed the EMU evaluation and that had at least one reported seizure during the EMU evaluation that was confirmed by triple review; (Investigator Reported Seizures + Triple Review).
Measure: Mean (95% Confidence Interval); unit: percentage of True Positive Detections
Groups:
- % Sensitivity: Total number of seizures detected by M106 divided by the total number of seizures reported (investigator + confirmation by triple review) during the EMU stay
Arm/Group | % Sensitivity
Number analyzed (Participants) | 18
percentage of True Positive Detections
  Ictal Tachycardia Seizures, SDA 2 (n=1; N=1) | 100 [NA to NA] — Confidence interval not computable where the mean sensitivity equals to 100%, or where number of patients within the setting is less than or equal to 2 (acceleration cannot be calculated).
  Ictal Tachycardia Seizures, SDA 4 (n=8; N=2) | 75 [NA to NA] — Confidence interval not computable where the mean sensitivity equals to 100%, or where number of patients within the setting is less than or equal to 2 (acceleration cannot be calculated).
  Ictal Tachycardia Seizures, SDA 6 (n=2; N=2) | 100 [NA to NA] — Confidence interval not computable where the mean sensitivity equals to 100%, or where number of patients within the setting is less than or equal to 2 (acceleration cannot be calculated).
  >= 70% heart rate increase, SDA 4 (n=3; N=2) | 66.7 [NA to NA] — Confidence interval not computable where the mean sensitivity equals to 100%, or where number of patients within the setting is less than or equal to 2 (acceleration cannot be calculated).
  >= 60% heart rate increase, SDA 2 (n=1; N=1) | 100 [NA to NA] — Confidence interval not computable where the mean sensitivity equals to 100%, or where number of patients within the setting is less than or equal to 2 (acceleration cannot be calculated).
  >= 60% heart rate increase, SDA 4 (n=4; N=2) | 50 [NA to NA] — Confidence interval not computable where the mean sensitivity equals to 100%, or where number of patients within the setting is less than or equal to 2 (acceleration cannot be calculated).
  >= 50% heart rate increase, SDA 4 (n=6; N=2) | 66.7 [NA to NA] — Confidence interval not computable where the mean sensitivity equals to 100%, or where number of patients within the setting is less than or equal to 2 (acceleration cannot be calculated).
  >= 50% heart rate increase, SDA 6 (n=1; N=1) | 100 [NA to NA] — Confidence interval not computable where the mean sensitivity equals to 100%, or where number of patients within the setting is less than or equal to 2 (acceleration cannot be calculated).
  >= 40% heart rate increase, SDA 4 (n=9; N=2)) | 66.7 [NA to NA] — Confidence interval not computable where the mean sensitivity equals to 100%, or where number of patients within the setting is less than or equal to 2 (acceleration cannot be calculated).
  >= 40% heart rate increase, SDA 6 (n=4; N=3)) | 100 [NA to NA] — Confidence interval not computable where the mean sensitivity equals to 100%, or where number of patients within the setting is less than or equal to 2 (acceleration cannot be calculated).
  >= 30% heart rate increase, SDA 6 (n=8; N=4)) | 100 [NA to NA] — Confidence interval not computable where the mean sensitivity equals to 100%, or where number of patients within the setting is less than or equal to 2 (acceleration cannot be calculated).
  >= 20% heart rate increase, SDA 6 (n=12; N=5) | 100 [NA to NA] — Confidence interval not computable where the mean sensitivity equals to 100%, or where number of patients within the setting is less than or equal to 2 (acceleration cannot be calculated).

3. Primary Outcome: Modeled Sensitivity Based on Heart Rate Increase Associated With Seizures by SDA Setting Post-Processed Through Bench-top Device Simulant
Description: Sensitivity is defined as the total number of seizures detected divided by the total number of seizures during the EMU stay. Data used to support sensitivity analyses included digital ECG/EEG files, corresponding M106 device downloads, and CRF data. Seizure onset times were compared with modeled M106 device detections at the least sensitive setting capable of detecting the seizure based on the corresponding change in heart rate. The participants' surface ECG data collected during the trial and passed through DMSDAT, a validated bench-top simulant of the Automatic Stimulation feature, was used to produce modeled results for each threshold for AutoStim setting (1;70%, 2;60%, 3;50%, 4;40%, 5;30% and 6;20%). Number of participants is total number of subjects who experienced seizures during the EMU stay.
  Bootstrap confidence intervals using 3000 bootstrap samples.
Time Frame: Epilepsy Monitoring Unit (EMU) Stay
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: percentage of True Positive Detections
Arm/Group | % Sensitivity
Number analyzed (Participants) | 18
percentage of True Positive Detections
  >= 70% heart rate increase at SDA 1 (n=5) | 100 [NA to NA] — Confidence interval left blank where the mean sensitivity equals to 100%
  >= 60% heart rate increase at SDA 2 (n=7) | 85.7 [70 to 100]
  >= 50% heart rate increase at SDA 3 (n=11) | 81.8 [57.14 to 100]
  >= 40% heart rate increase at SDA 4 (n=19) | 89.5 [73.68 to 100]
  >= 30% heart rate increase at SDA 5 (n=36) | 88.9 [76.67 to 97.37]
  >= 20% heart rate increase at SDA 6 (n=53) | 92.5 [79.66 to 100]

4. Primary Outcome: Potential False Positives Based on Heart Rate Increase Associated With Seizures by Randomized SDA Setting
Description: Potential false positive rate is defined as the sum across all patients of the total number of potential false positive detections divided by the sum across all patients of the appropriate monitoring time during the EMU stay. Data used to support the potential false positive rate analyses included digital ECG/EEG files retrieved from the EMU evaluation, corresponding M106 device downloads, and triple review results of EEG recordings.
  The evaluated EMU monitoring time includes a daily 3 minutes stepping exercise during which patients stepped up and down on a step stool at a submaximal effort leve.
Time Frame: Epilepsy Monitoring Unit (EMU) Stay
Population: ITT Population: all patients implanted with Model 106 VNS Therapy System Version 2 and who have any EMU record.
  10 participants analyzed for >=60% setting, 12 participants analyzed for >=40% setting, 8 participants analyzed for >=20% setting.
Measure: Number (95% Confidence Interval); unit: Potential False Positive per Hour
Groups:
- Potential False Positives: Potential False Positives Based on Heart Rate Increase Associated with Seizures by Randomized SDA Setting (AutoStim Per Hour)
Arm/Group | Potential False Positives
Number analyzed (Participants) | 30
Potential False Positive per Hour
  >=60%, SDA 2 | 0.5 [0.20 to 0.96]
  >=40%, SDA 4 | 2.7 [1.70 to 3.91]
  >=20%, SDA 6 | 7.2 [5.31 to 9.94]

5. Secondary Outcome: Validation of Cardiac R-Wave Detection
Description: Cardiac R-wave detection was evaluated against concurrent ECG data (i.e. detailed R-wave test) collected during implant, the first titration visit, at the beginning of the EMU stay, and at the 12 month visit. R-R intervals were calculated using detected R-waves from the Implantable Pulse Generator (IPG) and from a standard ECG monitor during a pre-specified time interval. A time series 10 seconds was recorded using the IPG SyncPulse feature. Simultaneously, a corresponding time series over the same interval was recorded using a standard ECG monitor. The total number of beats accurately detected in the entire study population is reported.
Time Frame: At Implant, First Titration Visit, Day 1 EMU and 12 Months
Population: ITT population
Measure: Number; unit: percentage of beats accurately detected
Groups:
- Beat Detection Sensitivity By Device IPG: Cardiac R-Wave Detection Sensitivity Based on Device IPG and ECG Monitor Comparison for 10 second Detection Window. "n" denotes the total number of patients with available R-R wave data at the visit time point.
Arm/Group | Beat Detection Sensitivity By Device IPG
Number analyzed (Participants) | 30
percentage of beats accurately detected
  At Implant (n=26) | 95.52
  First Titration Visit (n=19) | 98.74
  EMU Day 1 (n=29) | 99.71
  12 Month Follow-up (n=14) | 99.43

6. Secondary Outcome: Characterization of Latency Period: Analysis of Observed Latency for True Positive Detections by Randomized SDA Setting
Description: Latency is defined as the time difference between SDA detection time and the annotated seizure onset time. The earliest SDA detection was considered for each seizure. Seizure onset times were compared with M106 device detections at the randomized SDA setting. Negative latencies indicate that the SDA detection preceded the seizure onset time. The median latency is presented for seizures which met the definition of ictal tachycardia as well as all seizure types and indicate the observed latency range.
Time Frame: Epilepsy Monitoring Unit (EMU) Stay
Population: ITT Population n=total number of seizures in each category
Measure: Median (Full Range); unit: seconds
Groups:
- Latency Analysis of Ictal Tachycardia Seizures: The time difference between SDA detection of the ictal tachycardia seizure and the annotated seizure onset time.
  Ictal Tachycardia Seizure is defined as a seizure with an increase from a baseline heart rate to a rate that is greater than 100 bpm and is at least a 55% increase or 35 bpm.
- Latency Analysis of All Seizure Types: The time difference between SDA seizure detection time and the annotated seizure onset time (ALL seizures).
Arm/Group | Latency Analysis of Ictal Tachycardia Seizures | Latency Analysis of All Seizure Types
Number analyzed (Participants) | 30 | 30
seconds
  SDA 2 (n=1, 8) | 4 [4 to 4] | 19.5 [-89 to 92]
  SDA 4 (n=6,8) | 27.5 [12 to 57] | 27.5 [0 to 57]
  SDA 6 (n=2,37) | -14.5 [-42 to 13] | 7 [-112 to 110]

7. Secondary Outcome: Human Factors and Usability of the AspireSR® VNS Therapy® System.
Description: Usability survey data were collected from all site personnel who used the handheld programmer to evaluate the usability of the AspireSR® VNS Therapy® System.The device usability survey contained 17 questions that measure usability on a five-point Likert scale ranging from "Extremely Difficult" (5) to "Extremely Easy" (1). Site personnel were asked to assess usability of the software features, instructions for use, training materials, and overall usability of the system at four different time points. The time points include implant/recovery and the end of EMU.
  Usability was calculated as percentage of the users who found the usability of system to be "easy-2" or extremely easy-1".
Time Frame: At implant/recovery up to EMU Discharge (2 to 4 weeks)
Population: ITT Population
Measure: Number; unit: Percentage of participants rated 1 or 2
Groups:
- Implant/Recovery: Assessment of Device Usability at Implant and Recovery
- Day 5 EMU or EMU Discharge: Assessment of Device Usability at EMU (Day 5 or Discharge)
Arm/Group | Implant/Recovery | Day 5 EMU or EMU Discharge
Number analyzed (Participants) | 30 | 30
Percentage of participants rated 1 or 2
  Training Material (n=21, 23) | 76.2 | 73.9
  Physician's Manual (n=18, 20) | 61.1 | 70.0
  Laminated Instruction Card (n=20, 21) | 75.0 | 81.0
  Interrogation (Short) (n=22, 24) | 86.4 | 91.7
  Interrogation (Long) (n=21, 24) | 57.1 | 83.3
  Change Parameters (n=22, 24) | 90.9 | 95.8
  Heartbeat Sensitivity Configuration (n=20, 24) | 80.0 | 83.3
  Seizure Detection Configuration (n=21, 23) | 81.0 | 82.6
  System Diagnostic (n=21,24) | 85.7 | 87.5
  View Database (n=17, 22) | 58.8 | 72.7
  View Seizure Detection Data (n=15, 22) | 66.7 | 63.6
  Export Data (n=7, 15) | 100 | 66.7
  Generator Battery Status Indicators (n=20, 24) | 70.0 | 87.5
  Handheld Battery Status Indicator (n=19, 24) | 68.4 | 83.3
  Warning Messages (n=13, 24) | 84.6 | 87.5
  Overall Usability (n=20, 24) | 80.0 | 70.8

8. Secondary Outcome: Changes From Baseline in Seizure Frequency
Description: Seizure frequency was calculated at 3, 6, 12, 18 and 24 month follow-up visits based on seizure diary information and compared to baseline estimates. Response rate was computed and summarized for partial seizures (SPS, CPS and CPS with 2nd GTCs) and overall seizure types as the percentage of patients that achieved ≥50% seizure reduction per month from baseline by visit.
Time Frame: Up to 24 Month visit
Population: ITT population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Overall Seizure Responder Rate: Summary of Responders (>= 50% Seizure Counts Reduction per Month) by Visit (All seizure types)
- Partial Seizures: Summary of Responders (>= 50% Seizure Counts Reduction per Month) by Visit (Partial Seizures)
  Partial seizures consist of simple partial, complex partial, complex partial with secondarily generalized seizures.
Arm/Group | Overall Seizure Responder Rate | Partial Seizures
Number analyzed (Participants) | 30 | 30
Percentage of participants
  Follow-up 3 Month n=29,27 | 24.1 [10.30 to 43.54] | 25.9 [11.11 to 46.28]
  Follow-up 6 Month n=30,28 | 20.0 [7.71 to 38.57] | 25 [10.69 to 44.87]
  Follow-up 12 Month n=27,25 | 33.3 [16.52 to 53.96] | 36.0 [17.97 to 57.48]
  Follow-up 18 Month n=26,24 | 34.6 [17.21 to 55.67] | 37.5 [18.80 to 59.41]
  Follow-up 24 Month n=27,25 | 33.3 [16.52 to 53.96] | 36.0 [17.97 to 57.48]

9. Secondary Outcome: Changes in Seizure Severity Based on Physician Reported Questionnaire (NHS3)
Description: Investigators completed the National Hospital Seizure Severity Scale (NHS3) questionnaire at screening, at the end of the EMU stay (provided a seizure occurred during the EMU stay), and at follow-up visits. Severity was evaluated by seizure type. The range of NHS3 scale is 1-27 with 1 being the least severe and 27 being the most severe.
  Negative median value means improvement.
Time Frame: up to 24 Months Visit
Population: ITT Population
Measure: Median (Full Range); unit: Units on a scale
Groups:
- Simple Partial Seizures; Complex Partial Seizures (CPS); CPS w/2nd GTC; Generalized Tonic Clonic Sz: NHS3 Scores at Follow-Up Visits
Arm/Group | Simple Partial Seizures | Complex Partial Seizures (CPS) | CPS w/2nd GTC | Generalized Tonic Clonic Sz
Number analyzed (Participants) | 30 | 30 | 30 | 30
Units on a scale
  Baseline to EMU Discharge; n=11,19,5,3 | 0.00 [-4.0 to 1.0] | -1.00 [-10.0 to 0.0] | 0.00 [-14.0 to 0.0] | -4.00 [-5.0 to 0.0]
  Baseline to 3 Months; n=12,20,6,2 | 0.00 [-6.0 to 2.0] | -1.00 [-8.0 to 3.0] | 0.00 [-10.0 to 1.0] | -6.50 [-13.0 to 0.0]
  Baseline to 6 Months; n=9,20,5,3 | 0.00 [-2.0 to 9.0] | -1.33 [-9.0 to 3.2] | 0.00 [-14.0 to 0.0] | 0.00 [-12.0 to 9.0]
  Baseline to 12 Months; n=9,20,6,5 | 0.00 [-4.0 to 4.0] | -1.83 [-8.0 to 3.2] | 0.00 [-10.0 to 1.0] | -8.00 [-10.0 to 0.0]
  Baseline to 18 Months; n=7,20,7,3 | 2.00 [-3.0 to 6.0] | -1.50 [-12.0 to 5.0] | -1.0 [-8.0 to 1.0] | -7.00 [-10.0 to 0.0]
  Baseline to 24 Months; n=8,20,2,2 | -0.50 [-4.0 to 10.0] | -2.00 [-12.0 to 5.0] | -2.00 [-3.0 to -1.0] | -8.00 [-10.0 to -6.0]
Statistical Analysis 1: Comparison: Simple Partial Seizures; Baseline to EMU Discharge; Test type: Superiority or Other; p = 0.375, Signed Rank Test; Null hypothesis: change from the baseline is equal to zero. The alternative hypothesis: change from the baseline is not equal to zero
Statistical Analysis 2: Comparison: Simple Partial Seizures; Baseline to 3 Months; Test type: Superiority or Other; p = 0.156, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Simple Partial Seizures; Baseline to 6 months; Test type: Superiority or Other; p > 0.999, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: Simple Partial Seizures; Baseline to 12 Months; Test type: Superiority or Other; p = 0.906, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 5: Comparison: Simple Partial Seizures; Baseline to 18 Months; Test type: Superiority or Other; p = 0.188, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 6: Comparison: Simple Partial Seizures; Baseline to 24 Months; Test type: Superiority or Other; p = 0.906, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 7: Comparison: Complex Partial Seizures (CPS); Baseline to EMU Discharge; Test type: Superiority or Other; p < 0.001, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 8: Comparison: Complex Partial Seizures (CPS); Baseline to 3 Months; Test type: Superiority or Other; p = 0.106, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 9: Comparison: Complex Partial Seizures (CPS); Baseline to 6 Months; Test type: Superiority or Other; p = 0.012, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 10: Comparison: Complex Partial Seizures (CPS); Baseline to 12 Months; Test type: Superiority or Other; p = 0.008, s; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 11: Comparison: Complex Partial Seizures (CPS); Baseline to 18 Months; Test type: Superiority or Other; p = 0.009, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 12: Comparison: Complex Partial Seizures (CPS); Baseline to 24 Months; Test type: Superiority or Other; p = 0.029, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 13: Comparison: CPS w/2nd GTC; Baseline to EMU Discharge; Test type: Superiority or Other; p = 0.500, s; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 14: Comparison: CPS w/2nd GTC; Baseline to 3 Months; Test type: Superiority or Other; p > 0.999, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 15: Comparison: CPS w/2nd GTC; Baseline to 6 Months; Test type: Superiority or Other; p = 0.500, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 16: Comparison: CPS w/2nd GTC; Baseline to 12 Months; Test type: Superiority or Other; p = 0.500, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 17: Comparison: CPS w/2nd GTC; Baseline to 18 Months; Test type: Superiority or Other; p = 0.188, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 18: Comparison: CPS w/2nd GTC; Baseline to 24 Months; Test type: Superiority or Other; p = 0.500, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 19: Comparison: Generalized Tonic Clonic Sz; Baseline to EMU Discharge; Test type: Superiority or Other; p = 0.500, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 20: Comparison: Generalized Tonic Clonic Sz; Baseline to 3 Months; Test type: Superiority or Other; p > 0.999, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 21: Comparison: Generalized Tonic Clonic Sz; Baseline to 6 Months; Test type: Superiority or Other; p > 0.999, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 22: Comparison: Generalized Tonic Clonic Sz; Baseline to 12 Months; Test type: Superiority or Other; p = 0.125, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 23: Comparison: Generalized Tonic Clonic Sz; Baseline to 18 Months; Test type: Superiority or Other; p = 0.500, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 24: Comparison: Generalized Tonic Clonic Sz; Baseline to 24 Months; Test type: Superiority or Other; p = 0.500, Signed Rank Test; [statistical method as in outcome 9, analysis 1]

10. Secondary Outcome: Changes in Seizures Severity, Intensity & Post-Ictal Recovery Based on Patient Completed Seizure Severity Questionnaire (SSQ)
Description: Clinical outcomes such as seizure severity, intensity and post-ictal duration were also assessed during the long-term follow-up visits (3, 6, 12, 18 and 24 months) with patient reported questionnaires (SSQ; Seizure Severity Questionnaire). The range for SSQ (all sub-scores) is 1-7 with 1 being the least severe and 7 being the most severe.
  Mean SSQ scores at 3, 6, 12, 18 and 24 months were compared to baseline. A change from baseline is calculated as baseline minus follow-up visit score to correspond to the Minimally Important Change (MIC) criteria as defined in the Scoring Scheme for SSQ v2. Questionnaire. Subscale scores were averaged to compute the SSQ Total Score
Time Frame: Up to 24 Month visit
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- SSQ Scores at 3 Months; SSQ Scores at 6 Months; SSQ Scores at 12 Months; SSQ Scores at 18 Months; SSQ Scores at 24 Months: Change From Baseline at Each Category
Arm/Group | SSQ Scores at 3 Months | SSQ Scores at 6 Months | SSQ Scores at 12 Months | SSQ Scores at 18 Months | SSQ Scores at 24 Months
Number analyzed (Participants) | 30 | 30 | 30 | 30 | 30
Units on a scale
  SSQ Total Score n=24,27,26,23,20 MIC=0.48 | 0.516 (1.688) | 0.728 (1.567) | 0.354 (1.640) | 0.341 (1.461) | 0.966 (1.975)
  Activity During Seizure; n=26,28,27,25,22 MIC=0.50 | 1.115 (2.783) | 1.643 (2.714) | 0.907 (2.557) | 0.800 (2.441) | 1.818 (2.982)
  Overall Recovery; n=25,29,27,27,26 MIC=0.39 | 0.627 (3.101) | 0.663 (2.125) | 0.481 (2.514) | 0.280 (2.913) | 0.218 (2.783)
  Overall Severity; n=27,30,29,28,27 MIC=0.48 | 0.519 (3.022) | 0.589 (2.097) | 0.425 (2.486) | 0.131 (2.855) | 0.160 (2.806)
  Postictal Emotional Rec. n=26,29,28,27,26 MIC=0.42 | 0.397 (3.281) | 0.805 (2.832) | 0.179 (3.093) | -0.062 (3.480) | 0.359 (3.124)
  Postictal Physical Reco; n=27,30,28,28,27 MIC=0.34 | 0.975 (3.375) | 0.567 (2.208) | 0.393 (3.012) | 0.476 (3.018) | 0.012 (3.043)
  Postictal Cognitive Rec.;n=28,30,29,28,27 MIC=0.48 | 0.536 (3.467) | 0.578 (2.946) | 0.805 (2.814) | 0.274 (3.587) | 0.099 (3.404)
Statistical Analysis 1: Comparison: SSQ Scores at 3 Months; SSQ Total Score; Test type: Superiority or Other; p = 0.1529, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: SSQ Scores at 3 Months; Activity During Seizures Score; Test type: Superiority or Other; p = 0.0942, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: SSQ Scores at 3 Months; Overall Recovery Score; Test type: Superiority or Other; p = 0.2831, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: SSQ Scores at 3 Months; Overall Severity Score; Test type: Superiority or Other; p = 0.3639, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 5: Comparison: SSQ Scores at 3 Months; Postictal Emotional Recovery Score; Test type: Superiority or Other; p = 0.4470, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 6: Comparison: SSQ Scores at 3 Months; Postictal Physical Recovery Score; Test type: Superiority or Other; p = 0.1311, s; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 7: Comparison: SSQ Scores at 3 Months; Postictal Cognitive Recovery Score; Test type: Superiority or Other; p = 0.3898, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 8: Comparison: SSQ Scores at 6 Months; SSQ Total Score; Test type: Superiority or Other; p = 0.0511, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 9: Comparison: SSQ Scores at 6 Months; Activity During Seizures Score; Test type: Superiority or Other; p = 0.0019, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 10: Comparison: SSQ Scores at 6 Months; Overall Recovery Score; Test type: Superiority or Other; p = 0.1106, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 11: Comparison: SSQ Scores at 6 Months; Overall Severity Score; Test type: Superiority or Other; p = 0.1273, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 12: Comparison: SSQ Scores at 6 Months; Postictal Emotional Recovery Score; Test type: Superiority or Other; p = 0.1305, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 13: Comparison: SSQ Scores at 6 Months; Postictal Physical Recovery Score; Test type: Superiority or Other; p = 0.1123, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 14: Comparison: SSQ Scores at 6 Months; Postictal Cognitive Recovery Score; Test type: Superiority or Other; p = 0.2309, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 15: Comparison: SSQ Scores at 12 Months; SSQ Total Score; Test type: Superiority or Other; p = 0.3191, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 16: Comparison: SSQ Scores at 12 Months; Activity During Seizures Score; Test type: Superiority or Other; p = 0.0679, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 17: Comparison: SSQ Scores at 12 Months; Overall Recovery Score; Test type: Superiority or Other; p = 0.2082, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 18: Comparison: SSQ Scores at 12 Months; Overall Severity Score; Test type: Superiority or Other; p = 0.1790, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 19: Comparison: SSQ Scores at 12 Months; Postictal Emotional Recovery Score; Test type: Superiority or Other; p = 0.6869, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 20: Comparison: SSQ Scores at 12 Months; Postictal Physical Recovery Score; Test type: Superiority or Other; p = 0.6094, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 21: Comparison: SSQ Scores at 12 Months; Postictal Cognitive Recovery Score; Test type: Superiority or Other; p = 0.1530, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 22: Comparison: SSQ Scores at 18 Months; SSQ Total Score; Test type: Superiority or Other; p = 0.3339, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 23: Comparison: SSQ Scores at 18 Months; Activity During Seizures Score; Test type: Superiority or Other; p = 0.1473, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 24: Comparison: SSQ Scores at 18 Months; Overall Recovery Score; Test type: Superiority or Other; p = 0.5035, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 25: Comparison: SSQ Scores at 18 Months; Overall Severity Score; Test type: Superiority or Other; p = 0.6653, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 26: Comparison: SSQ Scores at 18 Months; Postictal Emotional Recovery Score; Test type: Superiority or Other; p = 0.8622, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 27: Comparison: SSQ Scores at 18 Months; Postictal Physical Recovery Score; Test type: Superiority or Other; p = 0.4456, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 28: Comparison: SSQ Scores at 18 Months; Postictal Cognitive Recovery Score; Test type: Superiority or Other; p = 0.6876, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 29: Comparison: SSQ Scores at 24 Months; SSQ Total Score; Test type: Superiority or Other; p = 0.0328, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 30: Comparison: SSQ Scores at 24 Months; Activity During Seizures Score; Test type: Superiority or Other; p = 0.0067, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 31: Comparison: SSQ Scores at 24 Months; Overall Recovery Score; Test type: Superiority or Other; p = 0.5928, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 32: Comparison: SSQ Scores at 24 Months; Overall Severity Score; Test type: Superiority or Other; p = 0.7179, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 33: Comparison: SSQ Scores at 24 Months; Postictal Emotional Recovery Score; Test type: Superiority or Other; p = 0.5014, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 34: Comparison: SSQ Scores at 24 Months; Postictal Physical Recovery Score; Test type: Superiority or Other; p = 0.9640, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 35: Comparison: SSQ Scores at 24 Months; Postictal Cognitive Recovery Score; Test type: Superiority or Other; p = 0.8537, Signed Rank Test; [statistical method as in outcome 9, analysis 1]

11. Secondary Outcome: Proportion of Seizures Ending During Stimulation by Type
Description: Clinical outcomes including seizure duration and cessation were assessed with vEEG during EMU stay. Number of seizures treated with Automatic Stimulation during EMU were evaluated. Of these seizures, those ending during the 60 second course of Automatic Stimulation were assessed and tabulated by seizure type.
Time Frame: Epilepsy Monitoring Unit (EMU) Stay
Population: ITT Population; All Treated Seizures n=total number of seizures
Measure: Number; unit: Percentage of Seizures Ending
Groups:
- Proportion of Seizures Ending During Stimulation by Type: EMU seizures that were treated with Automatic Stimulation and ended during the course of the stimulation
Arm/Group | Proportion of Seizures Ending During Stimulation by Type
Number analyzed (Participants) | 30
Percentage of Seizures Ending
  Overall (n=33) | 57.6
  Partial Seizures (not otherwise specified) (n=5) | 20
  Simple Partial Seizures (n=4) | 100
  Complex Partial Seizures (n=11) | 54.5
  Secondary Generalized Seizures (n=2) | 0.0
  Generalized Seizures (n=9) | 66.7
  Debilitating Seizures (CPS, SGS, GEN) (n=22) | 54.5
  Unknown Type (n=2) | 100

12. Secondary Outcome: Summary of Seizure Duration (Seconds) for All Seizure Types by Subgroup(ITT Population) (Only Seizures With Post Ictal Duration (Seconds) Annotated)
Description: Seizure duration was calculated using historical EEG data from patients enrolled in the trial and compared to the duration of seizures that occurred during the study EMU stay. The seizure start and end times were determined via clinical observation and/or through an adjudication process with qualified EEG reviewers.
Time Frame: Historical Seizures and Seizures during Epilepsy Monitoring Unit Stay
Population: Patients from the ITT population who had at least one seizure during the EMU stay and who had at least one historical seizure recorded (and duration was annotated). n=total number of seizures
Measure: Mean (Standard Deviation); unit: Seconds
Groups:
- Historical Seizures: Pre-study EEG recordings
- Terminated Seizures: Seizures which ended during Automatic Stimulation
- Unstimulated Seizures: Unstimulated seizures with >20% increase in heart rate.
Arm/Group | Historical Seizures | Terminated Seizures | Unstimulated Seizures
Number analyzed (Participants) | 30 | 30 | 30
Seconds
  Simple Partial Seizures n=6,4,0 | 45.5 (28.9) | 40.5 (32.1) | NA (NA) — no seizures reported
  Complex Partial Seizures n=60,6,7 | 150.2 (461.5) | 26.8 (16.2) | 150.7 (153.6)
  CPS Secondary Generalized n=12,0,0 | 107.3 (49.3) | NA (NA) — no seizures reported | NA (NA) — no seizures reported
  Generalized Seizures n=0,6,0 | NA (NA) — no seizures reported | 20.3 (10.4) | NA (NA) — no seizures reported
  Debilitating Seizures n=72,12,7 | 143.1 (421.5) | 23.6 (13.4) | 150.7 (153.6)

13. Secondary Outcome: Summary of Post Ictal Duration (Seconds) for All Seizure Types (ITT Population) (Only Seizures With Post Ictal Duration (Seconds) Annotated)
Description: Post-ictal duration was quantified by identifying the time at which the number of EEG channels within the 95% confidence interval of relative power reaches a number that is consistent with that during the pre-seizure period. This measure represents the amount of time required following a seizure until the EEG recovers to the pre-seizure state. It is used to objectively estimate patient recovery time. Historical seizures were baseline EEG recordings measured during monitoring prior to implantation. Post-ictal duration is only reported for seizures with Post Ictal Duration (seconds) annotated and >= 20% Heart Rate Rise
Time Frame: Historical Seizures and Seizures during Epilepsy Monitoring Unit Stay
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Historical Seizures | Terminated Seizures | Unstimulated Seizures
Number analyzed (Participants) | 30 | 30 | 30
Seconds
  Simple Partial Seizures n=5,4,0 | 274.6 (349.9) | 102.8 (110.2) | NA (NA) — No seizures recorded
  Complex Partial Seizures n=59,6,7 | 44.1 (67.3) | 85.7 (81.7) | 66.6 (99.9)
  CPS Secondary Generalized n=5,0,0 | 258.2 (199.3) | NA (NA) — No seizures recorded | NA (NA) — No seizures recorded
  Generalized Seizures n=0,1,0 | NA (NA) — No pre-study seizures (historical seizures) provided | 9.4 (0.0) | NA (NA) — No seizures recorded
  Debilitating Seizures n=64,7,7 | 60.9 (100.2) | 74.8 (79.9) | 66.6 (99.9)

14. Secondary Outcome: Changes in Quality of Life on Patient Reported Questionnaire (QOLIE-31-P)
Description: Quality of life data was collected using patient-completed QOLIE-31-P surveys and compared between baseline and follow-up visits. The MIC score for each subscale defines the threshold for Minimally Important Change. If a score exceeds the MIC Score, the improvement from baseline is considered clinically significant. The range for QOLIE-31-P (all sub-scores) is 0-100 with higher scores reflecting greater well-being.Subscale scores were averaged to compute the QOLIE Total Score.
Time Frame: up to 24 Months Visit
Population: ITT Population
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- QOLIE-31-P Scores at 3 Months; QOLIE-31-P Scores at 6 Months; QOLIE-31-P Scores at 12 Months; QOLIE-31-P Scores at 18 Months; QOLIE-31-P Scores at 24 Months: QOLIE-31-P Scores at Follow-Up Visits
Arm/Group | QOLIE-31-P Scores at 3 Months | QOLIE-31-P Scores at 6 Months | QOLIE-31-P Scores at 12 Months | QOLIE-31-P Scores at 18 Months | QOLIE-31-P Scores at 24 Months
Number analyzed (Participants) | 30 | 30 | 30 | 30 | 30
units on a scale
  QOLIE Overall Total (MIC=5.19) n=28,29,28,28,26 | 3.7 (16.6) | 4.4 (18.7) | 8.9 (18.4) | 10.2 (15.9) | 8.7 (25.3)
  Energy/Fatigue (MIC=5.25) n=28,29,28,28,25 | 2.3 (17.6) | -2.3 (17.9) | 4.3 (23.9) | 4.9 (21.0) | 6.9 (23.6)
  Emotional Well Being (MIC=4.76) n=28,29,28,28,26 | 0.4 (25.1) | -1.9 (21.4) | 7.1 (23.9) | 9.2 (24.7) | 8.2 (25.5)
  Social Functioning (MIC=3.95) n=27,28,26,27,26 | 11.7 (25.8) | 11.6 (26.3) | 20.1 (30.9) | 14.6 (18.6) | 10.2 (27.7)
  Cognitive functioning (MIC=5.34) n=28,29,28,27,26 | 1.3 (27.7) | 12.4 (37.7) | 8.4 (30.3) | 13.6 (30.4) | 9.6 (39.2)
  Medication Effects (MIC=5.00) n=28,29,28,26,26 | 4.5 (35.9) | 3.3 (27.5) | 0.9 (21.4) | 5.7 (31.1) | 1.1 (40.1)
  Seizure Worry (MIC=7.42) n=28,29,28,28,26 | 2.8 (26.6) | 2.1 (24.4) | 7.7 (27.9) | 8.1 (18.9) | 7.5 (31.0)
  Overall Quality of Life (MIC=6.42)n=28,29,28,28,26 | 3.7 (25.9) | 6.2 (25.4) | 14.9 (24.7) | 15.0 (23.1) | 16.0 (31.2)
Statistical Analysis 1: Comparison: QOLIE-31-P Scores at 3 Months; QOLIE Overall Total; Test type: Superiority or Other; p = 0.2079, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: QOLIE-31-P Scores at 3 Months; Energy/Fatigue Final Score; Test type: Superiority or Other; p = 0.6562, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: QOLIE-31-P Scores at 3 Months; Emotional well being Final Score; Test type: Superiority or Other; p = 0.9376, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: QOLIE-31-P Scores at 3 Months; Social Functioning Final Score; Test type: Superiority or Other; p = 0.0100, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 5: Comparison: QOLIE-31-P Scores at 3 Months; Cognitive functioning Final Score; Test type: Superiority or Other; p = 0.8532, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 6: Comparison: QOLIE-31-P Scores at 3 Months; Medication Effects Final Score; Test type: Superiority or Other; p = 0.4954, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 7: Comparison: QOLIE-31-P Scores at 3 Months; Seizure Worry Final Score; Test type: Superiority or Other; p = 0.1877, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 8: Comparison: QOLIE-31-P Scores at 3 Months; Overall Quality of Life Final Score; Test type: Superiority or Other; p = 0.4189, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 9: Comparison: QOLIE-31-P Scores at 6 Months; QOLIE Overall Total Score; Test type: Superiority or Other; p = 0.2365, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 10: Comparison: QOLIE-31-P Scores at 6 Months; Energy/Fatigue Final Score; Test type: Superiority or Other; p = 0.4138, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 11: Comparison: QOLIE-31-P Scores at 6 Months; Emotional well being Final Score; Test type: Superiority or Other; p = 0.8701, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 12: Comparison: QOLIE-31-P Scores at 6 Months; Social Functioning Final Score; Test type: Superiority or Other; p = 0.0527, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 13: Comparison: QOLIE-31-P Scores at 6 Months; Cognitive functioning Final Score; Test type: Superiority or Other; p = 0.1353, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 14: Comparison: QOLIE-31-P Scores at 6 Months; Medication Effects Final Score; Test type: Superiority or Other; p = 0.6927, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 15: Comparison: QOLIE-31-P Scores at 6 Months; Seizure Worry Final Score; Test type: Superiority or Other; p = 0.4964, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 16: Comparison: QOLIE-31-P Scores at 6 Months; Overall Quality of Life Final Score; Test type: Superiority or Other; p = 0.0238, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 17: Comparison: QOLIE-31-P Scores at 12 Months; QOLIE Overall Total Score; Test type: Superiority or Other; p = 0.0139, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 18: Comparison: QOLIE-31-P Scores at 12 Months; Energy/Fatigue Final Score; Test type: Superiority or Other; p = 0.2822, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 19: Comparison: QOLIE-31-P Scores at 12 Months; Emotional well being Final Score; Test type: Superiority or Other; p = 0.1363, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 20: Comparison: QOLIE-31-P Scores at 12 Months; Social Functioning Final Score; Test type: Superiority or Other; p = 0.0019, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 21: Comparison: QOLIE-31-P Scores at 12 Months; Cognitive functioning Final Score; Test type: Superiority or Other; p = 0.1293, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 22: Comparison: QOLIE-31-P Scores at 12 Months; Medication Effects Final Score; Test type: Superiority or Other; p = 0.5252, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 23: Comparison: QOLIE-31-P Scores at 12 Months; Seizure Worry Final Score; Test type: Superiority or Other; p = 0.0642, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 24: Comparison: QOLIE-31-P Scores at 12 Months; Overall Quality of Life Final Score; Test type: Superiority or Other; p = 0.0025, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 25: Comparison: QOLIE-31-P Scores at 18 Months; QOLIE Overall Total Score; Test type: Superiority or Other; p = 0.0024, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 26: Comparison: QOLIE-31-P Scores at 18 Months; Energy/Fatigue Final Score; Test type: Superiority or Other; p = 0.4464, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 27: Comparison: QOLIE-31-P Scores at 18 Months; Emotional well being Final Score; Test type: Superiority or Other; p = 0.0511, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 28: Comparison: QOLIE-31-P Scores at 18 Months; Social Functioning Final Score; Test type: Superiority or Other; p = 0.0002, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 29: Comparison: QOLIE-31-P Scores at 18 Months; Cognitive Functioning Final Score; Test type: Superiority or Other; p = 0.0296, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 30: Comparison: QOLIE-31-P Scores at 18 Months; Medication Effects Final Score; Test type: Superiority or Other; p = 0.3115, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 31: Comparison: QOLIE-31-P Scores at 18 Months; Seizure Worry Final Score; Test type: Superiority or Other; p = 0.0270, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 32: Comparison: QOLIE-31-P Scores at 18 Months; Overall Quality of Life Final Score; Test type: Superiority or Other; p = 0.0008, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 33: Comparison: QOLIE-31-P Scores at 24 Months; QOLIE Overall Total Score; Test type: Superiority or Other; p = 0.0683, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 34: Comparison: QOLIE-31-P Scores at 24 Months; Energy/Fatigue Final Score; Test type: Superiority or Other; p = 0.2226, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 35: Comparison: QOLIE-31-P Scores at 24 Months; Emotional well being Final Score; Test type: Superiority or Other; p = 0.0823, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 36: Comparison: QOLIE-31-P Scores at 24 Months; Social Functioning Final Score; Test type: Superiority or Other; p = 0.1459, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 37: Comparison: QOLIE-31-P Scores at 24 Months; Cognitive Functioning Final Score; Test type: Superiority or Other; p = 0.2610, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 38: Comparison: QOLIE-31-P Scores at 24 Months; Test type: Superiority or Other; p = 0.9119, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 39: Comparison: QOLIE-31-P Scores at 24 Months; Seizure Worry Final Score; Test type: Superiority or Other; p = 0.0826, Signed Rank Test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 40: Comparison: QOLIE-31-P Scores at 24 Months; Overall Quality of Life Final Score; Test type: Superiority or Other; p = 0.0036, Signed Rank Test; [statistical method as in outcome 9, analysis 1]

15. Secondary Outcome: Overall Summary of Seizure Intensity by Subgroup
Description: Quantitative evaluation of EEG was used to characterize the seizures that were treated with Automatic Stimulation. Intensity was evaluated by surveying the average power level from the 10-20 system EEG channel of maximum output during the course of the seizure. Intensity was only reported for seizures with intensity annotated and >= 20% Heart Rate Rise. The relative intensity was calculated by normalizing the power calculations to the pre-seizure state, and thus the reported changes are dimensionless. n= number of seizures
Time Frame: Historical Seizures and Seizures during Epilepsy Monitoing Unit Stay
Population: Patients from the ITT population who had at least one seizure during EMU stay and who had at least one historical seizure recorded. n=total number of seizures
Measure: Mean (Standard Deviation); unit: unitless
Groups:
- All EMU Stimulated Seizures: Stimulated Seizures with >= 20% increase in heart rate
- Unstimulated Seizures: Unstimulated seizures with =>20% increase in heart rate.
Arm/Group | Historical Seizures | All EMU Stimulated Seizures | Terminated Seizures | Unstimulated Seizures
Number analyzed (Participants) | 30 | 30 | 30 | 30
unitless
  Simple Partial Seizures n=6, 8, 4, 0 | 33.9 (33.9) | 225.3 (427.1) | 406.6 (581.0) | NA (NA) — no seizures recorded
  Complex Partial Seizures n=60, 9, 6, 7 | 205.4 (519.2) | 989.4 (2307.0) | 59.5 (65.2) | 51.6 (74.7)
  CPS Secondary generalized n=10, 2, 0, 0 | 435.1 (654.7) | 611.4 (832.2) | NA (NA) — no seizures recorded | NA (NA) — no seizures recorded
  Debilitating Seizures n=70, 12, 7, 7 | 238.2 (541.2) | 852.1 (2002.8) | 65.0 (61.3) | 51.6 (74.7)

16. Secondary Outcome: Post-stimulation Heart Rate Changes
Description: During a 1 hour period during the EMU stay, the VNS Therapy device was programmed to normal mode stimulation ON time 30 seconds, OFF time 5 minutes. AutoStim and Magnet Mode were programmed OFF. In this hour, 10 to 11 normal mode stimulations can be expected. Around each of these stimulations, ECG data were collected to assess potential stimulation related heart rate changes (during stimulation, after stimulation and after black-out time). A black-out time is a period after stimulation during which no seizure detections can occur, to ensure that potential stimulation related heart rate changes were not seen as ictal tachycardia that would trigger false positive detection. During the trial, the black-out time was programmed to 30 seconds. The heart rate changes for all stimulations and all patients were averaged.
Time Frame: EMU stay
Population: ITT population
Measure: Mean (Standard Deviation); unit: percentage change
Groups:
- Percentage Change in Heart Rate: Average percentage change in heart rate from pre-stimulation period to heart rate during VNS Therapy Stimulation, following VNS Therapy Stimulation, and following the black-out period.
Arm/Group | Percentage Change in Heart Rate
Number analyzed (Participants) | 30
percentage change
  During Stimulation | 0.74 (3.40)
  Post Stimulation | 0.09 (2.34)
  Post Black-Out time | -0.01 (2.92)

ADVERSE EVENTS:
Time Frame: From baseline up to 24 Months
Groups:
- VNS Therapy - Safety Population: All adverse events were collected from baseline up to the 24-month follow-up visit for all subjects treated/implanted with the AspireSR® VNS Therapy® system. All SAEs are reported in the SAE data table, whereas only the most common AEs (> 5%) are reported in the AE data table.
Arm/Group | VNS Therapy - Safety Population
Serious Adverse Events (participants affected / at risk) | 10/31
Other Adverse Events (participants affected / at risk) | 26/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VNS Therapy - Safety Population (N=31)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Hemorrhage Subcutaneous (Skin and subcutaneous tissue disorders) | 1 (1)
Convulsion (Nervous system disorders) | 3 (3)
Aphonia (Nervous system disorders) | 1 (1)
Status Epilepticus (Nervous system disorders) | 1 (1)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1)
Incision Site Pain (Injury, poisoning and procedural complications) | 1 (1)
Tibia Fracture (Injury, poisoning and procedural complications) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Tooth Abscess (Infections and infestations) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Psychotic Disorder (Psychiatric disorders) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VNS Therapy - Safety Population (N=31)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Dyspnea Exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Headache (Nervous system disorders) | 5 (5)
Dizziness (Nervous system disorders) | 3 (3)
Paresthesia (Nervous system disorders) | 2 (2)
Medical Device Pain (General disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Decreased Appetite (Metabolism and nutrition disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days